CLINICAL TRIAL: NCT04065113
Title: Middle Meningeal Artery (MMA) Embolization for Patients With Chronic Subdural Hematoma (cSDH)
Brief Title: Middle Meningeal Artery Embolization for Chronic Subdural Hematoma
Status: Withdrawn | Type: Observational
Why Stopped: due to reason 3 in the protocol- any new information becomes available during the trial that necessitates stopping the trial. New information became available with device no longer being investigational.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201905146
Record Dates: First submitted 2019-08-15; First posted 2019-08-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Chronic Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Polyvinyls; Ethanol; Polyvinyl Alcohol; Desmoglein 3; Craniotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Embolization Only: Medically managed patient receives middle meningeal artery embolization
  Interventions: Procedure: Middle Meningeal Artery Embolization with polyvinyl alcohol particles (PVA)
- Embolization + Evacuation: Participant receives standard of care evacuation and then undergoes MMA embolization
  Interventions: Procedure: Middle Meningeal Artery Embolization with polyvinyl alcohol particles (PVA); Procedure: Drainage of Subdural Hematoma
- Medical Management: Historical control of medically managed patients
- Surgical Patients: Historical control of patients receiving standard surgery alone
  Interventions: Procedure: Drainage of Subdural Hematoma

INTERVENTIONS:
Procedure: Middle Meningeal Artery Embolization with polyvinyl alcohol particles (PVA) — Seal off blood supply to the middle meningeal artery to prevent growth of subdural hematoma
  Other Names: MMA Embolization with polyvinyl alcohol (PVA) particles
  Groups: Embolization + Evacuation; Embolization Only
Procedure: Drainage of Subdural Hematoma — Drainage of subdural hematoma via burrhole or craniotomy
  Other Names: Burr Hole Drainage; Craniotomy
  Groups: Embolization + Evacuation; Surgical Patients

SUMMARY:
Endovascular middle meningeal artery (MMA) embolization is an emerging treatment for chronic subdural hematoma (cSDH). There is preliminary data to suggest that this minimally invasive therapy may be more efficacious and equally as safe compared to conventional, more invasive surgery. This study seeks to assess the safety and efficacy of middle meningeal artery embolization for chronic subdural hematoma as an adjunct to standard treatments, which include medical management and surgical evacuation.

DETAILED DESCRIPTION:
This study seeks to assess the safety and efficacy of middle meningeal artery embolization for chronic subdural hematoma in addition to standard treatments, which include close observation and surgical evacuation. Middle meningeal artery embolization has emerged recently as a minimally invasive and successful method of preventing re-accumulation of subdural hematoma, particularly for patients that are not obvious surgical candidates or those with recurrent or refractory hematomas. The outcomes of these two groups of patients who undergo middle meningeal artery embolization will be compared to matched historical controls.

Middle meningeal artery embolization is a minimally invasive angiography procedure completed with use of fluoroscopy. Access is obtained through the femoral or radial artery and a catheter is advanced to the MMA. Polyvinyl alcohol particles are then injected to seal off this portion of the artery and prevent any further blood flow into the subdural hematoma. Hemostasis is obtained at the access site and the patient is observed for 24-48 hours on a neurological care unit before discharge.

A head CT, NIHSS, and modified Rankin Score will be repeated on the following schedule: • Pre-Procedure

* 24 hours post procedure
* 7-10 days post procedure
* 30 days post procedure
* 90 days post procedure

Patients with chronic subdural hematoma undergo CT scans and neurologic assessments on hospital admission, as well as follow up CT scans and neurologic assessments to assess for any change in neurologic status or hematoma size. This study utilizes a standard of care follow up schedule to avoid exposing participants to extra radiation. Participants will be followed for study related purposes for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older undergoing treatment for a new diagnosis of chronic subdural hematoma (cSDH) or
* Patients 18 year or older who have undergone surgical evacuation of a subdural hematoma and have a significant residual hematoma status post-surgery or who develop a recurrent subdural hematoma.

and

* Minimal symptoms such as headache, altered mental status, or mild neurological deficit only
* Ability to understand and sign written informed consent by patient or LAR

Exclusion Criteria:

* Significant midline shift and/or neurologic symptoms requiring urgent decompression.
* Common carotid stenosis of over 50%.
* Significant contraindication to angiography (eg. kidney failure, difficult anatomy).
* SDH related to underlying condition
* Acute SDH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: number of participants reflects population with diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with recurrent or refractory hematoma (Radiographic resolution) | A head CT will be repeated 24 hours after the procedure, 7-10 days, 30 days, and 90 days post procedure to measure any change in size of the SDH compared to pre-procedure size
  The subdural hematoma persists or reoccurs
Number of patients requiring secondary evacuation surgery (Treatment Efficacy) | Evacuation surgery required within the 90 day follow up period
  The participant requires a post-procedure (post-MMA embolization) evacuation of the subdural hematoma due to re-occurrence or persistence of hematoma and symptoms

SECONDARY OUTCOMES:
Procedure-related complication rate (Safety) | Procedure-related complications will be compared between embolization and historical surgical patients assessed through study completion, 90 days
  Complication rate of embolization procedure vs surgery
Change in NIH Stroke Scale Score (Functional outcome) | Compared pre-procedure, 24 hours post-procedure, 7-10 days, 30 days, and 90 days post-procedure
  Change in score on National Institutes of Health Stroke Scale. The NIH Stroke Scale is used to quantify neurologic impairments. It consists of 11 items each scored between 0 and 4 points. The maximum score is 42, indicating severe impairment, and the minimum score is 0.
  Stroke severity 0 No stroke symptoms 1-4 Minor stroke 5-15 Moderate stroke 16-20 Moderate to severe stroke 21-42 Severe stroke
Change in modified Rankin Scale (Functional outcome) | Compared pre-procedure, 24 hours post-procedure, 7-10 days, 30 days, and 90 days post-procedure
  Change in score on modified Rankin Scale
  The modified Rankin Scale (mRS) measures the degree of disability or dependence after a stroke or other neurologic disease.
  The scale runs from 0-6, with 0 indicating perfect health with no symptoms to 6 indicating death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Change in size of subdural hematoma | Compared pre-procedure, 24 hours post-procedure, 7-10 days, 30 days, and 90 days post-procedure
  CT scan measurements of size of subdural hematoma

CONTACTS AND LOCATIONS:
Overall Officials: Joshua W Osbun, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT04065113/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT04065113/ICF_001.pdf